CLINICAL TRIAL: NCT05637307
Title: Sentinel NOSE Study: Prospective Registration Study on the Sentinel Node Procedure for Bulky Squamous Cell Carcinoma of the Nasal Vestibule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sentinel NOSE
Record Dates: First submitted 2020-11-19; First posted 2022-12-05 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Squamous Cell Carcinoma of the Nasal Vestibule
Keywords: nasal vestibule, sentinel node, nodal metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sentinel node procedure (Experimental): Participants will indergo the standard treatment for their disease ( i.e. brachytherapy) but a sentinel node procedure will be added to their treatment
  Interventions: Procedure: Sentinel node procedure

INTERVENTIONS:
Procedure: Sentinel node procedure — Injection of radio-active tracer in the tumor before brachytherapy treatment, visualization of sentinel nodes by SPECT, and extirpation of sentinel nodes by surgery

SUMMARY:
Management of the neck in Wang cT1-T2N0 nasal vestibule carcinoma (NVC) has been an ongoing point of discussion. As the disease is rare publications are scarce and published regional recurrence rates vary widely between 0% up to 23%. In general, literature recommends adequate radiological neck staging followed by a watchful waiting policy, as overall regional recurrence rates are low (5-10%).

However, according to recent findings, a subset of patients with large or voluminous cT1-T2N0 NVC is deemed at high risk of nodal involvement (20-40% regional recurrence) but receive no elective treatment, although it is well known that presence of nodal metastases impacts the prognosis of head and neck cancer (HNC) dramatically. Whereas elective neck dissection may be too aggressive, sentinel node biopsy (SNB) has been proven a reliable and safe alternative to bridge the gap between imaging and neck dissection.

SNB is currently routinely employed in most HNC centres in the Netherlands and is considered state of the art care, but its application in HNC is limited to oral cavity carcinoma and squamous cell carcinoma of the skin. Following the observation of increased risk of (occult) nodal metastases and regional recurrence in bulky tumors, the sentinel node procedure seems ideally suited for cT1-T2N0 NVC patients. Its superficial tumor localization is easily accessible for peritumoral Tc-99m-nanocolloid-ICG tracer injection. The purpose of this prospective registration study is to document the clinical introduction of the sentinel node procedure for bulky nasal vestibule carcinoma in our centre by protocol, and to identify and address possible unexpected difficulties specific for this tumor site. Ultimately, the goal will be routine and wide implementation of SNB in the NVC subgroup known to be at risk of nodal involvement, as a means to improve regional disease staging and control.

Objective: To prospectively document the introduction of the sentinel node procedure for bulky cT1-T2N0 nasal vestibule carcinoma in patients at risk of nodal involvement.

Study design: Single centre prospective registration study. To be extended with a second centre.

Study population: Patients with Wang cT1-T2N0 squamous cell carcinoma of the nasal vestibule, with tumor diameter ≥1.5 cm and/or tumor volume ≥1.5 cm3, with a WHO performance score of 2 or lower and no history of previous surgery or radiotherapy of the neck.

Interventions: 1. Subcutaneous peritumoral radioactive tracer injection followed by lymphoscintigraphy and Single Photon Emission Computed Tomography (SPECT) imaging for sentinel lymph node visualization.

2. Surgical sentinel node biopsy and histopathological examination of harvested nodes following the abovementioned imaging.

Main study parameters/endpoints: The primary endpoint of this study will be successful identification of sentinel nodes on lymphoscintigraphy and SPECT imaging. The procedure will be considered feasible when one or more sentinel nodes can be identified and localized in at least 7 out of the 10 patients..

DETAILED DESCRIPTION:
Management of the neck in Wang cT1-T2N0 nasal vestibule carcinoma (NVC) has been an ongoing point of discussion. As the disease is rare publications are scarce and published regional recurrence rates vary widely between 0% up to 23%. In general, literature recommends adequate radiological neck staging followed by a watchful waiting policy, as overall regional recurrence rates are low (5-10%).

However, according to recent findings, a subset of patients with large or voluminous cT1-T2N0 NVC is deemed at high risk of nodal involvement (20-40% regional recurrence) but receive no elective treatment, although it is well known that presence of nodal metastases impacts the prognosis of head and neck cancer (HNC) dramatically. Whereas elective neck dissection may be too aggressive, sentinel node biopsy (SNB) has been proven a reliable and safe alternative to bridge the gap between imaging and neck dissection.

SNB is currently routinely employed in most HNC centres in the Netherlands and is considered state of the art care, but its application in HNC is limited to oral cavity carcinoma and squamous cell carcinoma of the skin. Following the observation of increased risk of (occult) nodal metastases and regional recurrence in bulky tumors, the sentinel node procedure seems ideally suited for cT1-T2N0 NVC patients. Its superficial tumor localization is easily accessible for peritumoral Tc-99m-nanocolloid-ICG tracer injection. The purpose of this prospective registration study is to document the clinical introduction of the sentinel node procedure for bulky nasal vestibule carcinoma in our centre by protocol, and to identify and address possible unexpected difficulties specific for this tumor site. Ultimately, the goal will be routine and wide implementation of SNB in the NVC subgroup known to be at risk of nodal involvement, as a means to improve regional disease staging and control.

Objective: To prospectively document the introduction of the sentinel node procedure for bulky cT1-T2N0 nasal vestibule carcinoma in patients at risk of nodal involvement.

Study design: Single centre prospective registration study. To be extended with a second centre.

Study population: Patients with Wang cT1-T2N0 squamous cell carcinoma of the nasal vestibule, with tumor diameter ≥1.5 cm and/or tumor volume ≥1.5 cm3, with a WHO performance score of 2 or lower and no history of previous surgery or radiotherapy of the neck.

Interventions: 1. Subcutaneous peritumoral radioactive tracer injection followed by lymphoscintigraphy and Single Photon Emission Computed Tomography (SPECT) imaging for sentinel lymph node visualization.

2. Surgical sentinel node biopsy and histopathological examination of harvested nodes following the abovementioned imaging.

Main study parameters/endpoints: The primary endpoint of this study will be successful identification of sentinel nodes on lymphoscintigraphy and SPECT imaging. The procedure will be considered feasible when one or more sentinel nodes can be identified and localized in at least 7 out of the 10 patients..

The secondary outcomes will be: yield of at least one lymph node after biopsy, incidence of surgical complications and pain score during and after peritumoral tracer injection and tracer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* WHO performance score of 0, 1 or 2.
* Newly diagnosed T1 or T2 squamous cell carcinoma of the nasal vestibule.
* Tumor diameter ≥1.5 cm and/or tumor volume ≥1.5cm3
* Clinically negative neck (N0).
* Patients planned to undergo curative treatment.
* Patient provided written informed consent

Exclusion Criteria:

* Prior allergic reaction to either indocyanide green, 99m-Technetium nanocolloid or human colloidal albumin.
* Pregnancy.
* Previous surgery or radiotherapy of the neck.
* Concurrent secondary head-and-neck tumor.
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of identification of sentinel nodes | 1 week
  the number of identified nodes on SPECT that can actually be retrieved at subsequent surgery

SECONDARY OUTCOMES:
pain scores | 2 hours after injection
  Pain scores during and immediately after the injection of nanocolloid on a visual anlog scale ranging from 0-10
analgetics | 2 hours after injection
  use of analgetics ( both orally and locally administered)
surgical complications | 30 days after the procedure
  complications after surgery as registered in our hospital record database

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kaanders, Prof., PhD, MD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Anthoni van Leeuwenhoekhuis, Amsterdam
  - Radboud UMC, Nijmegen

IPD SHARING:
Plan to Share IPD: Yes
Data wil be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after closure of the study ( i.e.in 2 years time) for a time period of 5 years
Access Criteria: upon request